CLINICAL TRIAL: NCT00493792
Title: A Prospective, Randomized Study Comparing the Survival for X-3 Polyethylene to N2Vac Polyethylene When Used With the Triathlon Posterior Stabilized (PS) Total Knee System.
Brief Title: X-3 Polyethylene Survival Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Principal Investigator, Matthew P. Abdel, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-003093
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Results first posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Arthroplasty, Replacement, Knee; Total Knee Replacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (Active Comparator): Stryker Orthopaedics N2Vac Polyethylene when used with a Triathlon Posterior Stabilized total knee system. This is a fixed- bearing knee intended for use in patients undergoing cemented total knee arthroplasty.
  Interventions: Device: N2Vac Polyethylene
- Treatment (Experimental): Stryker Orthopaedics X3 Polyethylene when used with a Triathlon Posterior Stabilized total knee system. This is a fixed- bearing knee intended for use in patients undergoing cemented total knee arthroplasty.
  Interventions: Device: X3 Polyethylene

INTERVENTIONS:
Device: X3 Polyethylene — Highly cross-linked polyethylene (HXLPE).
  Other Names: X3
  Arms: Treatment
Device: N2Vac Polyethylene — Ultra-high-molecular-weight polyethylene (UHMWPE).
  Other Names: N2Vac
  Arms: Control

SUMMARY:
The goal of this clinical trial is to compare two types of polyethylene (Stryker Orthopaedics N2Vac and their X3 polyethylene) prostheses that are used in total knee replacements. The primary outcome will analyze whether or not prostheses require a revision surgery 10 years post knee replacement. Other outcomes such as reoperation rate, complications, radiographic results, and clinical outcomes will be collected.

It is hypothesized that X3 would perform equally well to N2Vac at 10 years.

DETAILED DESCRIPTION:
This is a prospective, randomized and blinded clinical trial. Participants will be assessed pre-operatively and post-operatively at three months and two, five, seven and ten years. The primary aim of the study is to compare the survivorship of two types of polyethylene (conventional N2Vac and highly cross-linked X3, both FDA approved via 510k clearance) used in a fixed-bearing total knee system in patients undergoing cemented total knee arthroplasty. Specifically, the primary endpoint will be the revision rate at ten years. These results will be measured through radiographs at each post-operative interval with an independent radiograph review being performed after all patients have reached 7 and 10 year follow-up. Secondary results will also be collected and will focus on disease-specific (Knee Society Scores), global (SF-12), and outcome measures. Radiographic results consisting of standing anteroposterior, lateral and Merchant views of the surgical knee will be recorded and analyzed. Completion of the initial investigation will occur at the 10-year interval after the last enrolled patient.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Subjects willing to sign the informed consent.
2. Subjects able to comply with follow-up requirements including post-operative weight bearing restrictions and self-evaluations.
3. Male and non-pregnant female subjects ages 21-85 years of age at the time of surgery.
4. Subjects requiring a primary total knee replacement.
5. Subjects with a diagnosis of osteoarthritis (OA), traumatic arthritis (TA), or avascular necrosis (AVN).
6. Subjects with intact collateral ligaments as determined by the surgeon investigator.

EXCLUSION CRITERIA:

1. Subjects with inflammatory arthritis.
2. Subjects with a history of total or unicompartmental reconstruction of the affected joint.
3. Subjects that have had a high tibial osteotomy or femoral osteotomy.
4. Subjects with neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
5. Subjects with a systemic or metabolic disorder leading to progressive bone deterioration.
6. Subjects that are immunologically compromised, or receiving chronic steroids (>30 days).
7. Subjects bone stock is compromised by disease or infection that cannot provide adequate support and/or fixation to the prosthesis.
8. Subjects with knee fusion to the affected joint.
9. Subjects with an active or suspected latent infection in or about the knee joint.
10. Subjects that are prisoners.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2007-02; Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Abdel, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at the following sites: Mayo Clinic in Rochester, MN, Mayo Clinic in Florida, and Mayo Clinic in Arizona. Patients, who met study criteria, planning to undergo a total knee replacement were offered study participation at their pre-operative visit.
Groups:
- Treatment: X3 Polyethylene when used with a Triathlon Posterior Stabilized total knee system. This is a fixed- bearing knee intended for use in patients undergoing cemented total knee arthroplasty.
  Stryker X3 Crosslink Polyethylene: Highly cross-linked polyethylene (HXLPE).
Period: Overall Study
Arm/Group | Control | Treatment
Started | 254 | 264
Year 2 | 245 | 256
Year 5 | 233 | 241
Year 7 | 207 | 211
Completed (Participants who had study data available at the 10 year post-operation mark.) | 163 | 163
Not Completed | 91 | 101
Not completed — Death | 55 | 50
Not completed — Lost to Follow Up or Lack of Efficacy | 36 | 51

BASELINE CHARACTERISTICS:
Population: Patients were recruited from three academic, tertiary-care referral centers within one healthcare network. Patients approached for enrollment received a primary unilateral TKA for a diagnosis of osteoarthritis (OA), avascular necrosis (AVN) or posttraumatic arthritis. Patients were randomized into the control or treatment group. A Modified Intent-to-Treat (MITT) population was used.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Treatment | Total
Number analyzed (Participants) | 254 | 264 | 518
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9) | 67 (9) | 67 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 155 | 300
  Male | 109 | 109 | 218
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 169 (10) | 169 (10) | 169 (10)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 92 (21) | 92 (21) | 92 (21)
BMI, kg/m^2 [Mean (Standard Deviation); unit: Kilogram-Square Meter (kg/m^2)] | 32 (7) | 32 (6) | 32 (7)
Previous knee surgery, n (%) [Count of Participants; unit: Participants]
  Yes, previous knee surgery | 91 | 82 | 173
  No, previous knee surgery | 157 | 179 | 336
  Unknown | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Prosthesis Survivorship Free of Revision
Description: The survival of prostheses free of revision 10 years post operation.
Time Frame: From operation to 10 years post-operative
Population: Patients were recruited from three academic, tertiary-care referral centers within one healthcare network. Patients approached for enrollment received a primary unilateral total knee arthroplasty (TKA) for a diagnosis of osteoarthritis (OA), avascular necrosis (AVN) or posttraumatic arthritis.
Measure: Number (95% Confidence Interval); unit: percentage of prosthesis survivorship
Groups:
- Treatment: Stryker Orthopaedics X3 Polyethylene when used with a Triathlon Posterior Stabilized total knee system. This is a fixed- bearing knee intended for use in patients undergoing cemented total knee arthroplasty.
  X3 Crosslink Polyethylene: Highly cross-linked polyethylene (HXLPE).
Arm/Group | Control | Treatment
Number analyzed (Participants) | 254 | 264
percentage of prosthesis survivorship | 96 [93 to 98] | 97 [94 to 99]
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.47, Regression, Cox; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.29 to 1.77]

2. Secondary Outcome: Prosthesis Survivorship Free of Reoperation
Description: The survival of prostheses free of reoperation 10 years post operation.
Time Frame: From operation to 10 years post-operative
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of prosthesis survivorship
Arm/Group | Control | Treatment
Number analyzed (Participants) | 254 | 264
percentage of prosthesis survivorship | 92 [89 to 96] | 96 [93 to 99]
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.06, Regression, Cox; Hazard Ratio (HR) = .49, 95% CI 2-sided [0.23 to 1.03]

3. Secondary Outcome: Prosthesis Survivorship Free of Complications
Description: The survival of prostheses free of related complications (non-operative) 10 years post operation.
Time Frame: From operation to 10 years post-operative
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of prosthesis survivorship
Arm/Group | Control | Treatment
Number analyzed (Participants) | 254 | 264
percentage of prosthesis survivorship | 84.9 [80.2 to 89.5] | 88.8 [84.5 to 92.8]
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.193, Regression, Cox; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [.45 to 1.18]

4. Secondary Outcome: Knee Society Score (KSS)
Description: The KSS evaluates pain, stability and range of motion. The scale ranges between scores of 0-100. The maximum score of 100 points is reached when there is no pain, with good alignment of the knee in extension, and at least 125° of range of motion, without any anteroposterior or mediolateral instability. Deductions are made for flexion contracture, loss of extension and poor alignment. Higher scores indicate better knee conditions, while lower scores indicate worse knee conditions.
Time Frame: Pre-operative (baseline) and 10-years post-operative
Population: Patients who completed the Knee Society Score at baseline and patients who completed the Knee Society Score at 10-years post-operation.
  Data was not collected nor analyzed for 90 patients in the control arm, and 93 patients in the treatment arm at the 10 year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 123 | 121
score on a scale
  Baseline Score | 39.9 (14.19) | 39.0 (12.56)
  10-Year Follow-Up Score: number analyzed (Participants) | 33 | 28
  10-Year Follow-Up Score | 77.6 (8.60) | 76.5 (6.32)

5. Secondary Outcome: Knee Society Score (KSS): Function
Description: The Function KSS evaluates the walking distance and the act of climbing and descending stairs. The scale ranges between 0-100. The maximum score of 100 points is attributed to the individual capable of walking unlimited distances without walking aids, and of climbing and descending stairs normally. Deductions are made for the use of canes, crutches or walking frame. Higher scores indicate better knee conditions, while lower scores indicate worse knee conditions.
Time Frame: Pre-operative (baseline) and 10-years post-operative
Population: Patients who completed the Knee Society Function Score at baseline and patients who completed the Knee Society Function Score at 10-years post-operation.
  Data was not collected nor analyzed for 62 patients in the control arm, and 47 patients in the treatment arm at the 10 year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 156 | 159
score on a scale
  Baseline Score | 58.3 (17.38) | 59.1 (15.48)
  10-Year Follow-Up Score: number analyzed (Participants) | 94 | 112
  10-Year Follow-Up Score | 70.2 (26.25) | 70.3 (26.16)

6. Secondary Outcome: 12-Item Short Form Health Survey (SF-12): Mental Health Score
Description: The SF-12 questionnaire uses questions selected from the longer SF-36 Health Survey to measure patient wellness and quality of life. The scoring algorithm is calibrated so that an average healthy person would have a t-score of 50 points with a standard deviation of 10. Higher scores indicate better mental health.
Time Frame: Pre-operative (baseline) and 10-years post-operative
Population: Patients who completed the SF-12 Mental Health Score at baseline and patients who completed the SF-12 Mental Health Score at 10-years post-operation.
  Data was not collected nor analyzed for 187 patients in the control arm, and 193 patients in the treatment arm at the 10 year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 228 | 233
score on a scale
  Baseline Score | 56 (9.64) | 56.2 (8.89)
  10-Year Follow-Up Score: number analyzed (Participants) | 41 | 40
  10-Year Follow-Up Score | 56.8 (6) | 56.3 (7.65)

7. Secondary Outcome: 12-Item Short Form Health Survey (SF-12): Physical Health Score
Description: The SF-12 questionnaire uses questions selected from the longer SF-36 Health Survey to measure patient wellness and quality of life. The scoring algorithm is calibrated so that an average healthy person would have a t-score of 50 points with a standard deviation of 10. Higher scores indicate better physical health.
Time Frame: Pre-operative (baseline) and 10-years post-operative
Population: Patients who completed the SF-12 Physical Health Score at baseline and patients who completed the SF-12 Physical Health Score at 10-years post-operation.
  Data was not collected nor analyzed for 187 patients in the control arm, and 193 patients in the treatment arm at the 10 year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 228 | 233
score on a scale
  Baseline Score | 32.5 (8.34) | 33.2 (8.59)
  10-Year Follow-Up Score: number analyzed (Participants) | 41 | 40
  10-Year Follow-Up Score | 41.9 (11.28) | 44.4 (10.37)

8. Secondary Outcome: Comparison of Radiographic Success/Failure Between Groups
Description: Radiographic review for success and or failure of the TKA prostheses at 10 years post-operation. A migrating or shifting prosthesis with or without the disappearance of radiolucent lines is considered a failure.
Time Frame: 10 years post-operative
Population: Patients who completed 10-year post-operation radiographs of the study-related prosthetic joint.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 40 | 23
Participants
  Loosening and/or Osteolysis | 0 | 0
  Tibial component bone-cement interface: Non-progressive radiolucent lines | 7 | 2
  Femoral component bone-prosthesis interface: Radiolucent lines | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored post-operatively day 1 until study completion (10 years).
Arm/Group | Control | Treatment
All-Cause Mortality (participants affected / at risk) | 55/254 | 50/264
Serious Adverse Events (participants affected / at risk) | 0/254 | 0/264
Other Adverse Events (participants affected / at risk) | 0/254 | 0/264

LIMITATIONS AND CAVEATS:
Wear related failures require significant lengths of time in which to present, longer-term data are necessary to definitively uncover differential wear and osteolysis risk between HXLPE and UHMWPE. The present investigation strictly utilized cemented femoral and tibial component fixation and posterior stabilized bearing designs. Additionally, 14% of patients were lost to follow-up by 10 years with the potential for bias therein; however, there was no differential attrition between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-04-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT00493792/Prot_SAP_000.pdf